CLINICAL TRIAL: NCT01915810
Title: Using Physical Activity to Facilitate Smoking Cessation Among African American Adults
Brief Title: Physical Activity in Promoting Smoking Cessation in African Americans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-0183; NCI-2015-01057 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0183 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Current Smoker; Healthy Subject
MeSH Terms: interventions — Tobacco Use Cessation Devices; Nicotine

ARMS (3):
- Arm I (pre-quit physical activity) (Experimental): Participants receive telephone-based cessation counseling over 15-20 minutes 1-2 weeks before assigned quit date and nicotine patch for 6 weeks. Beginning 2 weeks before the assigned quit date, participants receive a Walking Program guide and engage in the SCwPA comprising brisk, self-paced walking with a goal of 150 minutes of exercise activity per week for 5 weeks.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Drug: Nicotine Patch; Other: Questionnaire Administration; Other: Tobacco Cessation Counseling
- Arm II (quit day physical activity) (Experimental): Participants receive telephone-based cessation counseling over 15-20 minutes 1-2 weeks before assigned quit date and nicotine patch for 6 weeks. Beginning on the assigned quit date, participants receive a Walking Program guide and engage in the SCwPA comprising brisk, self-paced walking with a goal of 150 minutes of exercise per week for 5 weeks.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Drug: Nicotine Patch; Other: Questionnaire Administration; Other: Tobacco Cessation Counseling
- Arm III (no physical activity) (Active Comparator): Participants quit smoking on an assigned date and receive telephone-based cessation counseling over 15-20 minutes 1-2 weeks before assigned quit date and nicotine patch for 6 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nicotine Patch; Other: Questionnaire Administration; Other: Tobacco Cessation Counseling

INTERVENTIONS:
Behavioral: Exercise Intervention — Complete SCwPA intervention
  Arms: Arm I (pre-quit physical activity); Arm II (quit day physical activity)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nicotine Patch — Receive nicotine patch
  Other Names: NicoDerm CQ; Nicotine Skin Patch; Nicotine Transdermal Patch
Other: Questionnaire Administration — Ancillary studies
Other: Tobacco Cessation Counseling — Receive smoking cessation counseling

SUMMARY:
This randomized pilot clinical trial studies the use of physical activity in promoting the discontinuation of the habit of smoking (smoking cessation) in African Americans. Participating in physical activity during an actual smoking quit attempt may work better in helping African Americans stop smoking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of a Smoking Cessation with Physical Activity (SCwPA) intervention among an African American (AA) church-based sample of adult current smokers.

II. Conduct post-intervention focus groups to obtain feedback from pilot participants regarding the acceptability of the SCwPA project design and procedures.

III. Examine how physical activity (PA) and the timing of PA initiation affects the mechanisms underlying cessation among an AA church-based sample of adult daily smokers who are attempting to quit.

OUTLINE: Participants are randomized to 1 of 3 arms.

ARM I (PRE-QUIT PHYSICAL ACTIVITY): Participants receive telephone-based cessation counseling over 15-20 minutes 1-2 weeks before assigned quit date and nicotine patch for 6 weeks. Beginning 2 weeks before the assigned quit date, participants receive a Walking Program guide and engage in the SCwPA comprising brisk, self-paced walking with a goal of 150 minutes of exercise activity per week for 5 weeks.

ARM II (QUIT DAY PHYSICAL ACTIVITY): Participants receive telephone-based cessation counseling over 15-20 minutes 1-2 weeks before assigned quit date and nicotine patch for 6 weeks. Beginning on the assigned quit date, participants receive a Walking Program guide and engage in the SCwPA comprising brisk, self-paced walking with a goal of 150 minutes of exercise per week for 5 weeks.

ARM III (NO PHYSICAL ACTIVITY): Participants quit smoking on an assigned date and receive telephone-based cessation counseling over 15-20 minutes 1-2 weeks before assigned quit date and nicotine patch for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported African-American race
* Current daily smoker (has smoked >= 100 cigarettes in lifetime per self-report, smoked >= 5 cigarettes per day for the last 6 months per self-report)
* Self-reports motivation to quit smoking within the next 2 weeks
* Reports willingness to engage in a physical activity-based smoking cessation intervention
* Has a home address and a functioning home and/or cell phone number
* Able to engage in moderate intensity physical activity as determined by the Physical Activity Readiness Questionnaire (PAR-Q) or by physicians clearance (letter from physician or nurse practitioner) if currently taking medication for blood pressure or diabetes
* Willingness to wear the nicotine patches provided in the study as recommended
* Have an expired carbon monoxide (CO) level > 8 parts per million (ppm) suggestive of current smoking
* Blood pressure =< 140/90mm or by physicians clearance (letter from physician or nurse practitioner) if blood pressure reading > 140/90mm Hg

Exclusion Criteria:

* Contraindication for nicotine patch use
* Regular use of tobacco products other than cigarettes in the last 30 days (including black & milds)
* Current or planned future use of any nicotine replacement or pharmacological product for smoking cessation other than the study patches
* Pregnancy or lactation
* Another household member enrolled in the study
* A schedule not accommodating to the study procedures, or unwillingness to adhere to the procedures

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-01-29 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility, defined as >= 75% of eligible/screened participants choose to enroll in the study | Up to 8 weeks
Retention feasibility, defined as an overall retention rate of 80% and if each enrolled participant completes >= 66.7% of study visits (>= 6 of 9 study visits) | Up to 8 weeks
Post intervention focus group analysis | Up to 8 weeks
  Each focus group will use a semi-structured interview guide for consistency, which will consist of approximately 15 open-ended questions. If results do not suggest intervention feasibility, post-intervention focus groups will help to identify why feasibility was not achieved. Focus group transcripts will be imported into a qualitative data analysis software program, such as NVivo, to facilitate data retrieval and analysis and to organize data by themes based on phrases, patterns, relationships, and commonalties or disparities.

SECONDARY OUTCOMES:
Mechanisms underlying smoking cessation (e.g., stress, positive and negative affect, depression, smoking urges, self-efficacy, motivation, PA enjoyment, and heart rate variability) | Up to 8 weeks
  Validated questionnaires via associated scoring manuals or by convention in the literature will be scored. Descriptive statistics, including mean and variance estimates with 95% confidence intervals, relevant to each of the identified mechanism variables, for each intervention group will be generated. Group*time effects with regard to stress, positive and negative affect, depression, smoking urges, self-efficacy, motivation, and heart rate variability will be examined using repeated measure analyses of variance as the primary analysis technique.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna McNeill, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org